CLINICAL TRIAL: NCT02794935
Title: The Effects of Inspiratory Muscle Training in Patients With Heart Failure and Obstructive Sleep Apnea Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Cruz Alta (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado do Rio Grande do Sul, Brazil (Other); Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CAAE: 25471413.7.0000.5322
Record Dates: First submitted 2016-05-31; First posted 2016-06-09 (Estimated); Last update posted 2016-08-09 (Estimated); Status verified 2016-08

CONDITIONS: Chronic Heart Failure
Keywords: inspiratory muscle training; heart failure; obstructive sleep apnea
MeSH Terms: conditions — Heart Failure; Sleep Apnea, Obstructive

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Inspiratory muscle training (IMT) (Experimental): Participants will be submitted to a linear pressure resistance (PowerBreathe) with an inspiratory load of 30% of maximal inspiratory pressure (adjusted weekly), seven days a week, session duration of 30 minutes for 12 weeks. During training, participants will be instructed to maintain diaphragmatic breathing with a breathing rate of 15-20 cycles/min. Inspiratory load will be set at 30% of maximum static inspiratory pressure, and weekly training loads will be adjusted to maintain 30% of MIP. Each week, six training sessions will be held at home and a training session will be supervised in the research center.
  Interventions: Other: Inspiratory muscle training (IMT)
- Sham IMT (Placebo Comparator): Participants will be submitted to inspiratory muscle training with the same equipment as the intervention group, but without a load generating resistance. Sham IMT Participants will receive IMT for 30 min, 7 times per week for 12 weeks using Inspiratory muscle trainer device (PowerBreathe). During training, participants will be instructed to maintain diaphragmatic breathing with a breathing rate of 15-20 cycles/min, but without a load generating resistance. Each week, six training sessions will be held at home and a training session will be supervised in the research center.
  Interventions: Other: Sham IMT

INTERVENTIONS:
Other: Inspiratory muscle training (IMT) — Participants will be submitted to a linear pressure resistance (PowerBreathe) with an inspiratory load of 30% of maximal inspiratory pressure (adjusted weekly), seven days a week, session duration of 30 minutes for 12 weeks. During training, participants will be instructed to maintain diaphragmatic breathing with a breathing rate of 15-20 cycles/min. Inspiratory load will be set at 30% of maximum static inspiratory pressure, and weekly training loads will be adjusted to maintain 30% of MIP. Each week, six training sessions will be held at home and a training session will be supervised in the research center.
  Arms: Inspiratory muscle training (IMT)
Other: Sham IMT — Participants will be submitted to inspiratory muscle training with the same equipment as the intervention group, but without a load generating resistance. Sham IMT Participants will receive IMT for 30 min, 7 times per week for 12 weeks using Inspiratory muscle trainer device (PowerBreathe). During training, participants will be instructed to maintain diaphragmatic breathing with a breathing rate of 15-20 cycles/min, but without a load generating resistance. Each week, six training sessions will be held at home and a training session will be supervised in the research center
  Arms: Sham IMT

SUMMARY:
This research aims to evaluate the effects of inspiratory muscle training (IMT) on apnea hypopnea index, sleepiness, sleep quality, cognitive function, motor task, executive function, quality of life, chemoreflex sensitivity and vagal modulation of heart rate in patients with heart failure and obstructive sleep apnea syndrome.

DETAILED DESCRIPTION:
Patients with heart failure will be selected through the Outpatient of the Rio Grande do Sul, for convenience. Subsequently, patients will be subjected to test respiratory muscle strength (manometer), respiratory muscle endurance, portable polysomnography, sleepiness, sleep quality, cognitive function (mini-mental state examination), motor task (execution of a sequence of digital movements), executive function, quality of life (SF-36), maximum exercise testing, chemoreflex sensitivity (peripheral chemoreflex by transient hypoxia and central chemoreflex by hypercapnic hyperoxia) and vagal modulation of heart rate (spectral analysis) before the start of the training protocol. Patients will be randomized to inspiratory muscle training or control group. Inspiratory muscle training will be performed for 30 minutes a day, 7 days a week, for 12 weeks with muscle training device (PowerBreathe). There will be a weekly monitoring in the Clinical Research Center of the institution where the maximal inspiratory pressure (MIP) and respiratory training techniques will be reassessed and readjusted (30% of MIP). The control group will be submitted to respiratory training techniques with muscle training device (PowerBreathe) without load. After this period, all initial tests will be reassessed. A group study with 15 heart failure patients without obstructive sleep apnea syndrome will be included.

ELIGIBILITY:
Inclusion Criteria:

* Heart failure patients with obstructive sleep apnea- hypopnea
* Heart failure patients without sleep apnea
* Left ventricle fraction ejection < 51 % for men and < 53% for woman
* Must be clinically stable
* New York Heart Association I, II and III
* Without changes in medication for the last three months.

Exclusion Criteria:

* Unstable angina
* Atrial fibrillation
* Acute myocardial infarction (<6 months)
* Recent heart surgery (<6 months)
* Chronic metabolic disease
* Infectious disease
* Anemia
* Severe hypoxemia
* Neuromuscular disease
* Diabetes mellitus
* Obesity
* Use of continuous positive airway pressure
* Smoking
* Pulmonary disease (forced vital capacity <80% of predicted and / or forced expiratory volume in one second <70% predicted).

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2016-06; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Apnea hypopnea index | 12 weeks
  measured by portable polysomnography [in events/hour]

SECONDARY OUTCOMES:
sleepiness | 12 weeks
  measured by Epworth Sleepiness Scale [in score]
sleep quality | 12 weeks
  assessed by the Pittsburgh sleep quality index [in score]
cognitive function | 12 weeks
  measured by the mini-mental state [in points]
motor task | 12 weeks
  assessed by the execution of a sequence of digital movements [in time required and number of execution errors]
executive function measured by Trail Making Test | 12 weeks
  measured by Trail Making Test. In Part A, participants are asked to link numbered points randomly distributed on a sheet of paper in ascending order according to numbers. In Part B, the participants are asked to link numbers and letters alternately [in time of test performance, counts the number of errors, and calculates the difference in times: B-A.].
quality of life assessed by the The Medical Outcomes Study - Short-form 36 (SF-36) | 12 weeks
  assessed by the The Medical Outcomes Study - Short-form 36 (SF-36)
peak oxygen consumption | 12 weeks
  It will be assessed using of treadmill stress test with Bruce protocol. The peak oxygen consumption will be estimated according to the method established by the American College Sports Medicine [in mL.kg-1.min-1]
chemoreflex sensitivity | 12 weeks
  peripheral chemoreflex will be assessed by transient hypoxia [in L.min-1.mmHg] and central chemoreflex by hypercapnic hyperoxic in [L. min-1. %SatO2]
vagal modulation measured by heart rate monitoring in the time domain (spectral analysis) | 12 weeks
  measured by heart rate monitoring in the time domain by spectral analysis [in normalized units]

CONTACTS AND LOCATIONS:
Overall Officials: Carine C Callegaro, PhD, Principal Investigator — University of Cruz Alta
Locations (1):
- University of Cruz Alta, Cruz Alta, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: Yes
The volunteers will receive the results of the evaluations pre and post-intervention by the of the study.